CLINICAL TRIAL: NCT03114904
Title: Comparison of the Efficacy of a Protocol for the Withdrawal of Neurosedation From the Usual Strategy in Cerebroses: Randomized Controlled Trial.
Brief Title: Comparison of the Efficacy of a Protocol for the Withdrawal of Neurosedation From the Usual Strategy in Cerebroses
Acronym: NEUROSEV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: PI2015_843_0019
Record Dates: First submitted 2017-04-04; First posted 2017-04-14 (Actual); Last update posted 2020-07-20 (Actual); Status verified 2020-07

CONDITIONS: Withdrawal Syndrome; Cerebral Lesion
MeSH Terms: conditions — Substance Withdrawal Syndrome

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- "Usual" weaning management (Other)
  Interventions: Other: Variation of Jasinski score between H0 (stop of sedatives) and H6
- Introduction to H2 for the discontinuation of therapeutics (Other)
  Interventions: Other: Variation of Jasinski score between H0 (stop of sedatives) and H6

INTERVENTIONS:
Other: Variation of Jasinski score between H0 (stop of sedatives) and H6 — To compare the effectiveness of a withdrawal management protocol with the usual management in cerebral patients (Subarachnoid haemorrhage (HSA), stroke and head trauma (CT))

SUMMARY:
The withdrawal syndrome in benzodiazepines and morphine is common in intensive care, the incidence is estimated at 32.1%.

Cerebrospatized patients are probably more prone to withdrawal because they require high doses of sedation.

Moreover, this syndrome is probably deleterious on the cerebral hemodynamics (high point of the therapeutic management).

ELIGIBILITY:
Inclusion Criteria:

* Major Patient
* Admitted in Neuroreanimation
* Cerebroséé (TC-HSA-AVC)
* Mono or multi failing
* After a neurosedation ≥ 3 days by hypnotic type benzodiazepine (Midazolam®) and morphinomimetic (Sufentanyl®) in IVSE
* Affiliation to Social Security
* Agreement of the person of confidence

Exclusion Criteria:

* Addiction to opiates, cocaine or cannabis
* Neurological Pathology Before Hospitalization
* Patient suffering from cardiac arrest
* Pregnant woman
* Sedation window
* Patient under tutelage or curatorship or deprived of public law

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2016-02-27 (Actual); Primary Completion 2018-05-16 (Actual); Study Completion 2018-05-16 (Actual)

PRIMARY OUTCOMES:
A variation of the Jasinski score between H0 (stop sedation) and H6. This score measures the signs of withdrawal | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens Picardie, Amiens, Picardie, France